CLINICAL TRIAL: NCT07403175
Title: Synergistic Impact of Postural Correction Interventions and Sustained Natural Apophyseal Glides on Severity, Disability and Quality of Life in Patients With Migraine
Brief Title: Synergistic Impact of Postural Correction Interventions and Sustained Natural Apophyseal Glides in Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/01104
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Migraine
Keywords: Disability; Headache; Migraine; Sustained Natural Apophyseal Glide; Neck Disability
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sustained Natural Apophyseal Glides & Postural Correction Exercises (Experimental)
  Interventions: Other: Sustained Natural Apophyseal Glides; Other: Postural Correction Exercises; Other: Conventional Physical Therapy
- Sustained Natural Apophyseal Glides (Active Comparator)
  Interventions: Other: Sustained Natural Apophyseal Glides; Other: Conventional Physical Therapy

INTERVENTIONS:
Other: Sustained Natural Apophyseal Glides — Headache SNAG: A posteroanterior mobilization of the second cervical vertebrae is maintained for 10-30 seconds having the patient comfortably seated on a chair or couch. A maximum of six repetitions were administered. The patient is administered SNAG mobilization by placing the medial border of the thumb's distal phalanx on the spine of one vertebra above while standing behind the patient. The thumb tips were positioned at a 45° angle, and another thumb is used to provide the glides. Glides are performed in 3 sets and 6 times during the session.
  Reverse Headache SNAG: Anterio-posterior mobilization of the second cervical vertebrae is maintained for 10-30 seconds having the patient comfortably seated on a chair or couch. A maximum of 6 repetitions were administered.
  Other Names: SNAGs
Other: Postural Correction Exercises — The main exercises used in this group are stretching, strengthening, and endurance exercise to maintain a healthy posture and correct the faulty posture due to weakened and tightened muscles Each subject will receive 6 treatment sessions spread over 4 consecutive weeks and each treatment session will not extend beyond 30 min.
  * Stretching exercises
  * Levator scapulae stretching
  * Upper trapezius stretching
  * Scalenes muscle stretching
  * Pectoralis major stretch
  * Pectoralis minor stretch
  * Sternocleidomastoid stretch
  * Strengthening Exercises
  * Lower trapezius strengthening
  * Rhomboids strengthening
  * Deep cervical flexors strengthening
  * Endurance Training
  Arms: Sustained Natural Apophyseal Glides & Postural Correction Exercises
Other: Conventional Physical Therapy — * Hot pack for 20 minutes on the neck region (upper trapezius) in sitting position.
  * Soft tissue mobilization includes deep tissue massage locally to the cervical region by applying pressure with fingers and palms.
  * Isometrics of neck in which the patient is seated on a chair or standing, or in a comfortable position having spine in a neutral position. Placing hands on patient's forehead by asking the patient to gently push head forward while simultaneously resisting the movement therapist's hands. Hold the contraction for 5-10 seconds, then relax. this movement was repeated in all directions.

SUMMARY:
This study was conducted to evaluate the synergistic impact of postural correction interventions and sustained natural apophyseal glides on severity, quality of life and disability in patients with migraine.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of episodic migraine made by the primary investigator according to ICHD-2.
* Symptoms must include at least two of the following: Unilateral pain, Pulsating/throbbing pain, Nausea, Vomiting, Photophobia/phonophobia.
* Participants should be full time employees or Desktop users.
* Participants have a history of at least migraine >4 days per month.
* Participants having history of migraine lasting from 4-72 hours
* Age group between 22 and 45 years.
* Both gender male and female.
* Participants who agree to cut-off any pharmacological treatment during study.
* Participants should have an average score between 3-6 on pain intensity scale.

Exclusion Criteria:

* Participants having active migraine and other headache types e.g. Cluster headache.
* Previous neck/head trauma from >2 years.
* Any neck/head surgery >2 years
* Spinal infections/diseases e.g. Tumor, TB spine
* Any history of neurological disorders e.g. stroke, abcess, haemorrhage, haematoma
* Severe Osteoporosis
* Pregnancy
* Upper motor neuron disease, cervical stenosis, and metabolic diseases in bone and joint.
* Ongoing radiotherapy, chemotherapy, steroid therapy, or anticoagulants.
* Psychiatric diseases such as phobia/obsession and depression.

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | From enrollment to the end of treatment at 4 weeks.
  The NRS is used to gauge the patient's degree of pain. On a 0-10 scale, where 0 represents no pain, 1-3 represents mild pain, 4-6 represents moderate pain, and 7-10 represents severe pain, this tool is frequently used to gauge the intensity of pain. Patients rate how much pain they are currently experiencing as well as how much pain they have experienced in the past 24 hours. The patient's level of pain might be represented by the average of three evaluations or by any single value
Migraine Specific Quality of Life Questionnaire (MSQ Version 2.1) | From enrollment to the end of treatment at 4 weeks.
  This questionnaire is used to evaluate migraine patient's quality of life. The 14-item MSQ version 2.1 measures QOL impacts in three domains: Role function-restrictive (RFR), which measures the functional impact of migraine through limitations on daily social and work activities; Role function-preventive (RFP), which measures the impact of migraine through prevention of daily work and social activities; and Emotional function (EF), which measures the emotional impact of migraine through three items. The raw total score was the sum of all item scores, which were rescaled from 0 to 100, with a higher score denoting better quality of life. Raw scores in each domain were calculated as the sum of all item scores.
Migraine Disability Assessment Scale (MDA) | From enrollment to the end of treatment at 4 weeks.
  The Migraine Disability Assessment Scale (MIDAS) is intended to assist individuals and medical professionals in comprehending how migraines affect day-to-day living. MIDAS gives a more accurate view of the overall impact of migraines by evaluating how frequently they occur and how they interfere with social activities, employment, and domestic duties. It is simpler to customize therapy to meet each patient's needs when the information is used to determine treatment choices and monitor progress overtime. In the end, it's a tool that facilitates improved communication and assistance in migraine management by allowing patients to share their experiences and difficulties.

SECONDARY OUTCOMES:
ROM Cervical Spine (Flexion) | From enrollment to the end of treatment at 4 weeks.
  Changes in cervical spine flexion ROM at baseline and 4th week of intervention was measured using goniometer.
ROM Cervical Spine (Extension) | From enrollment to the end of treatment at 4 weeks.
  Changes in cervical spine extension ROM at baseline and 4th week of intervention was measured using goniometer.
ROM Cervical Spine (Lateral Flexion) Left Side | From enrollment to the end of treatment at 4 weeks.
  Changes in cervical spine lateral flexion on left side ROM at baseline and 4th week of intervention was measured using goniometer.
ROM Cervical Spine (Lateral Flexion) Right Side | From enrollment to the end of treatment at 4 weeks.
  Changes in cervical spine lateral flexion on right side ROM at baseline and 4th week of intervention was measured using goniometer.
ROM Cervical Spine (Rotation) Left Side | From enrollment to the end of treatment at 4 weeks.
  Changes in cervical spine rotation on left side ROM at baseline and 4th week of intervention was measured using goniometer.
ROM Cervical Spine (Rotation) Right Side | From enrollment to the end of treatment at 4 weeks.
  Changes in cervical spine rotation on right side ROM at baseline and 4th week of intervention was measured using goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Rafia Mannan, MS-SPT, Principal Investigator — Riphah International University
Locations (1):
- Abdul Ahaad Hospital, Sialkot, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No